CLINICAL TRIAL: NCT07172529
Title: Evaluation of Pulmonary Function, Respiratory Muscle Strength, Peripheral Muscle Strength and Functional Capacity in Individuals Undergoing Minimally Invasive Cardiac Surgery
Brief Title: Pulmonary Function, Muscle Strength, and Functional Capacity in Minimally Invasive Cardiac Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Zehra Can Karahan (Other)
Responsible Party: Sponsor-Investigator, Zehra Can Karahan, Asst. Prof., Atılım University
Organization: Atılım University (Other)
Other Study IDs: 3dcd45b218264a9a
Record Dates: First submitted 2025-08-18; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Muscle Weakness | Patient; Pulmonary Function; Functional Capacity
Keywords: cardiac surgery; muscle weakness; pulmonary function; kinesiophobia; functional capacity
MeSH Terms: conditions — Muscle Weakness; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate pulmonary function, respiratory muscle strength, peripheral muscle strength, and functional capacity in adult patients undergoing either minimally invasive cardiac surgery (via mini-thoracotomy) or conventional sternotomy for coronary artery bypass grafting (CABG) at Gülhane Training and Research Hospital.The main questions it aims to answer are:

Does minimally invasive cardiac surgery preserve pulmonary function better than conventional sternotomy? Does minimally invasive cardiac surgery result in less respiratory and peripheral muscle weakness compared to conventional sternotomy? Researchers will compare patients undergoing minimally invasive surgery with those undergoing conventional sternotomy to determine differences in pulmonary function, respiratory muscle strength, peripheral muscle strength, and functional capacity.

Participants will:

Undergo preoperative and postoperative (day 4) assessments including spirometry, inspiratory/expiratory mouth pressure measurements, and peripheral muscle strength testing (handgrip, shoulder flexion/abduction, hip flexion, knee extension).

Perform functional capacity tests (30-second sit-to-stand test, 6-minute walk test).

Complete questionnaires assessing pain (McGill Pain Questionnaire) and fear of movement (Tampa Scale of Kinesiophobia).

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is one of the most commonly performed surgical procedures for patients with complex coronary artery disease. While the standard approach is through median sternotomy, minimally invasive cardiac surgery performed via mini-thoracotomy has gained popularity due to potential benefits such as smaller incisions, reduced surgical trauma, lower risk of sternal complications, shorter hospital stays, and faster mobilization. However, its effects on pulmonary function, respiratory muscle strength, peripheral muscle strength, and functional capacity have not been sufficiently clarified.

Postoperative pulmonary complications are a significant concern in cardiac surgery. Procedures involving cardiopulmonary bypass may result in atelectasis, pneumonia, pleural effusion, phrenic nerve injury, and diaphragm dysfunction. These complications can impair respiratory mechanics, delay rehabilitation, and increase morbidity and mortality. Therefore, identifying surgical approaches that better preserve pulmonary and muscular function is of great clinical importance.

This observational study will prospectively evaluate adult patients undergoing CABG at Gülhane Training and Research Hospital, comparing two groups: those receiving minimally invasive cardiac surgery via mini-thoracotomy and those undergoing conventional sternotomy. The primary outcomes are changes in pulmonary function parameters measured by spirometry (FVC, FEV1, PEF) from baseline to postoperative day 4. Secondary outcomes include respiratory muscle strength (MIP, MEP), peripheral muscle strength (handgrip, shoulder flexion/abduction, hip flexion, knee extension), functional capacity (30-second sit-to-stand test, 6-minute walk test), pain intensity (McGill Pain Questionnaire), and fear of movement (Tampa Scale of Kinesiophobia).

All assessments will be performed twice: before surgery (preoperative baseline) and on postoperative day 4. This time frame was chosen to capture early postoperative functional changes, which may influence short-term recovery and rehabilitation strategies. By comparing the two surgical techniques, this study aims to determine whether minimally invasive cardiac surgery provides better preservation of pulmonary and muscular function, ultimately supporting improved patient-centered outcomes and guiding clinical decision-making in surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* Scheduled for elective cardiac surgery via either minimally invasive approach (mini-thoracotomy) or conventional sternotomy at Gülhane Training and Research Hospital
* Able to provide written informed consent

Exclusion Criteria:

* Previous history of cardiac surgery
* Presence of orthopedic or neurological disorders affecting mobility or muscle strength
* Postoperative cerebrovascular event
* Requirement for mechanical ventilation > 24 hours postoperatively
* Intensive care unit stay > 48 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-80 years) scheduled for elective coronary artery bypass grafting at Gülhane Training and Research Hospital, either via minimally invasive mini-thoracotomy or conventional sternotomy approach.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Function - Forced Vital Capacity (FVC) | Baseline [preoperative] and postoperative day 4)
  Forced Vital Capacity measured by spirometry. Results will be reported in liters (L).
Change in Pulmonary Function - Forced Expiratory Volume in 1 second (FEV1) | Baseline to postoperative day 4
  Forced Expiratory Volume in 1 second measured by spirometry. Results will be reported in liters (L).
Change in Respiratory Muscle Strength - Maximal Inspiratory Pressure (MIP) | Baseline [preoperative] and postoperative day 4
  Inspiratory muscle strength measured with mouth pressure device. Results will be reported in cmH₂O.
Change in Respiratory Muscle Strength - Maximal Expiratory Pressure (MEP) | Baseline [preoperative] and postoperative day 4
  Expiratory muscle strength measured with mouth pressure device. Results will be reported in cmH₂O.
Change in Handgrip Strength | Baseline to postoperative day 4
  Handgrip strength measured with handheld dynamometer. Results will be reported in kilograms (kg).
Change in Knee Extension Strength | Baseline to postoperative day 4
  Knee extension strength measured with handheld dynamometer. Results will be reported in kilograms (kg).
Change in Functional Capacity - 30-Second Sit-to-Stand Test | Baseline to postoperative day 4
  Number of repetitions performed during the 30-second sit-to-stand test. Results will be reported as number of repetitions.
Change in Functional Capacity - 6-Minute Walk Distance | Baseline to postoperative day 4
  Distance covered during the 6-minute walk test. Results will be reported in meters (m).

SECONDARY OUTCOMES:
Change in Pain Intensity - McGill Pain Questionnaire | Baseline and postoperative day 4
  Pain intensity assessed with the McGill Pain Questionnaire. Results will be reported as score values (units on a scale). Minimum score: 0 (no pain) Maximum score: 78 (maximum pain intensity) Higher scores indicate worse pain.
Change in Kinesiophobia - Tampa Scale of Kinesiophobia (TSK-17) | Baseline and postoperative day 4
  Fear of movement assessed with the Tampa Scale of Kinesiophobia (TSK-17). Results will be reported as score values ranging from 17 to 68 (units on a scale).Higher scores indicate greater fear of movement (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Can Karahan, PHD, Study Director — Atılım University
Locations (1):
- Atilim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT07172529/Prot_SAP_000.pdf